CLINICAL TRIAL: NCT04117646
Title: Validity of the French Version of the Child's Chronic Rhinosinusitis Questionnaire
Acronym: SN5-FR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190791; ID RCB : 2019-A00387-50 (Other: ANSM)
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis
Keywords: Chronic rhinosinusitis of children; Sinus and nasal quality of life survey questionnaire (SN-5); Translation in French of the SN-5
MeSH Terms: conditions — Fistula | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients of 2 and 12 years of age with chronic rhinosinusitis.
  Interventions: Other: Sinus and nasal quality of life survey questionnaire (SN-5)
- Controls: Subjects of 2 and 12 years of age without chronic rhinosinusitis.
  Interventions: Other: Sinus and nasal quality of life survey questionnaire (SN-5)

INTERVENTIONS:
Other: Sinus and nasal quality of life survey questionnaire (SN-5) — Subjects respond to the translated questionnaire twice at 15 days apart.
  Other Names: Patient questionnaire

SUMMARY:
A single quality questionnaire evaluating the symptoms of chronic rhinosinusitis in children currently exists. It has been validated in English for children aged 2 to 12. It comprises five areas of quality of life, each rated by a score ranging from 1 to 7 : sinus infection, nasal obstruction, allergic symptoms, emotional distress and activity limitation, coupled with an overall assessment of quality of life with an analogue visual scale (score from 1 to 10). This SN-5 (sinus and nasal quality of life survey) score showed excellent statistics of reproducibility, internal validity and ease of response. It is currently used in several international publications evaluating chronic sinus pathology in children.

The objective of the study is to validate the translation of the SN-5 questionnaire in French.

DETAILED DESCRIPTION:
Chronic rhinosinusitis is a common pathology that entrains significant medical consumption. The prevalence of chronic rhinosinusitis in children is estimated to be 7.6%. Cardinal symptoms include nasal congestion, purulent rhinorrhea, facial pain, and persistent daytime cough. All these nasal symptoms often have an impact on the quality of life. The main objective of medical treatment is to improve this quality of life.

The treatment of chronic rhinosinusitis is mainly medical and includes nose washes with physiological serum, topical or general corticosteroid treatment or antibiotics. Surgical treatments such as adenoidectomy or endonasal functional surgery are reserved for medical treatment failures. According to a European consensus paper of 2012, the surgical strategy of the chronic rhinosinusitis of the child must start with a adenoidectomy with physiological serum washes, and then secondarily a endonasal functional surgery.

The ability of quality of life questionnaires to measure subjective symptoms over a certain length of time can help in the medical decision by determining the benefit of taking care. A single quality questionnaire evaluating the symptoms of chronic rhinosinusitis in children currently exists. It has been validated in English for children aged 2 to 12. It comprises five areas of quality of life, each rated by a score ranging from 1 to 7 : sinus infection, nasal obstruction, allergic symptoms, emotional distress and activity limitation, coupled with an overall assessment of quality of life with an analogue visual scale (score from 1 to 10). This SN-5 (sinus and nasal quality of life survey) score showed excellent statistics of reproducibility, internal validity and ease of response. It is currently used in several international publications evaluating chronic sinus pathology in children.

The objective of the study is to validate the translation of the SN-5 questionnaire in French.

ELIGIBILITY:
Inclusion Criteria:

* Non-opposition of the holders of parental authority and the subject to participation in the study
* Subjects between 2 and 12 years of age Patients : - Patients followed in consultation at Necker Hospital in pediatric department of otolaryngology and cervico-facial surgery for chronic rhinosinusitis (rhinosinusitis more than 12 weeks)

Controls :

- Subject without chronic rhinosinusitis at the time of inclusion and without chronic rhinitis history

Exclusion Criteria:

French language not spoken by parents

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients followed by the department of otolaryngology and cervico-facial surgery of Necker-Enfants Malades hospital and siblings for the control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Reproducibility | 1 year
  Reproducibility of the questionnaire completed by a subject at 15 days apart. Student t-test.
Consistency reliability test | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.
Item-total Pearson correlation | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.
Principal components analysis | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Leboulanger, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gargula S, Luscan R, Drummond D, Denoyelle F, Couloigner V, Leboulanger N, Simon F. French translation and validation of the Sinus and Nasal Quality of Life Survey (SN-5) in children. Int J Pediatr Otorhinolaryngol. 2021 Jun;145:110706. doi: 10.1016/j.ijporl.2021.110706. Epub 2021 Apr 6. PMID 33862327